CLINICAL TRIAL: NCT00422526
Title: Randomised Study to Examine the Effectiveness of Progesterone in Preventing Severe Preterm Delivery
Brief Title: Progesterone for Prevention of Preterm Birth in Women With Short Cervix: Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 03WH13
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Last update posted 2007-01-17 (Estimated); Status verified 2007-01

CONDITIONS: Preterm Birth; Pregnancy Trimester, Second
Keywords: Preterm delivery, short cervix, progesterone
MeSH Terms: conditions — Premature Birth; Neoplasm Metastasis | interventions — Utrogestan

INTERVENTIONS:
Drug: Micronised progesterone (Utrogestan)

SUMMARY:
The aim of our study is to evaluate the effect of use of prophylactic vaginal progesterone on the incidence of severe preterm delivery, defined as delivery before 33+6 weeks in women with a short cervical length of 15mm.

DETAILED DESCRIPTION:
BACKGROUND The results of randomized studies have shown that the prophylactic use of progesterone in women who previously delivered prematurely reduces the risk of recurrence. Asymptomatic women found to have a short cervix (< 15 mm) at mid-gestation are at greatly increased risk for spontaneous early preterm delivery and it is uncertain whether in such women the risk is reduced by progesterone.

METHODS Cervical length was measured by transvaginal sonography at 22 (range 20-25) weeks in 24,620 pregnant women attending for routine antenatal care. The cervix was 15 mm or less in 413 (1.7%), and 250 (60.5%) of these women participated in a randomized study of vaginal progesterone (200 mg per night) vs identical-looking placebo, between 24 and 34 weeks. Primary outcome was the frequency of spontaneous delivery before 34 weeks (238 days) of pregnancy. Analysis was performed according to the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* All women with singleton or twin pregnancies attending for routine ultrasound examination at 20-25 weeks of gestation with a short cervical length (<15 mm).

Exclusion Criteria:

* Women with major fetal abnormalities,
* Painful regular uterine contractions, or history of ruptured membranes or cervical cerclage in-situ were excluded from screening.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250
Dates: Start 2003-09; Study Completion 2006-11

PRIMARY OUTCOMES:
Spontaneous delivery before 34 completed weeks (238 days) of gestation.

SECONDARY OUTCOMES:
Birth weight, fetal or neonatal death, major adverse outcome before discharge from hospital and need for neonatal special care (admission to special care baby unit, phototherapy, treatment of proven or suspected sepsis, or blood transfusion).

CONTACTS AND LOCATIONS:
Overall Officials: Kypros H Nicolaides, MD, PhD, Principal Investigator — King's College London
Locations (8):
- Hospital do Servidor Publico Estadual-FMO, São Paulo, São Paulo, Brazil
- Hospital Clinico Universidad de Chile, Santiago, Santiago Metropolitan, Chile
- University Hospital, Larissa, Larissa, Greece
- United Kingdom (5):
  - University Hospital of Lewisham, London, London
  - Queen Elizabeth Hospital, NHS Trust Woolwich, London, London
  - King's College Hospital NHS Foumdation Trust, London, London
  - Southend University Hospital, Essex, London, London
  - Darent Valley Hospital, Kent

REFERENCES:
- [Derived] Fonseca EB, Celik E, Parra M, Singh M, Nicolaides KH; Fetal Medicine Foundation Second Trimester Screening Group. Progesterone and the risk of preterm birth among women with a short cervix. N Engl J Med. 2007 Aug 2;357(5):462-9. doi: 10.1056/NEJMoa067815. PMID 17671254